CLINICAL TRIAL: NCT03792230
Title: Comparison Of The Effects Of Different Body Mechanics Education Methods On Pain, Disability And Quality Of Life: Randomised Controlled Study
Brief Title: Comparison Of The Effects Of Different Body Mechanics Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Ozgu Bakcek, Master of Science, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ozgubakcek
Record Dates: First submitted 2018-12-30; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Nursing Care; Patient Education
Keywords: Lumbar disc hernia surgery; Body mechanics; Patient education; Quality of life; Disability; Pain; Nursing
MeSH Terms: conditions — Pain | interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: prospective randomised controlled study
Who Masked: Investigator
Masking Description: Because of only one investigator, there is no blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video (Experimental): This group received educatıon via video material
  Interventions: Behavioral: Video
- Brochure (Experimental): This group received education via written material (brochure)
  Interventions: Behavioral: Brochure
- Control (No Intervention): This group received standart clinical education

INTERVENTIONS:
Behavioral: Video — Video group receive body mechanic education via CD material,
  Arms: Video
Behavioral: Brochure — Brochure group receive body mechanic education via written material (brochure)
  Arms: Brochure

SUMMARY:
The study evaluated the comparison of the different patient education methods. The study involved two stages of data collection: one during the preoperative period, the other during the sixth postoperative week.

DETAILED DESCRIPTION:
Before commencing the study, we informed participants who met the inclusion criteria about the scope of the study and obtained their written and oral consent. Participants in each group completed the data collection form regarding patients' characteristics, the SF-MPQ, the ODI and the Physical Functioning and Bodily Pain subscales of the SF-36. A day before LDH (Lumbar Disc Hernia) surgery, participants in the control group received standard clinical education, whereas ones in the intervention groups received either video- or brochure-based education. Participants in the brochure group learned about the proper use of body mechanics from the "Body Mechanics Educational Brochure for LDH Patients" and demonstrations performed by primary investigator after which we answered any questions that participants asked. Brochure-based education took nearly 15 min, and participants could keep the brochures after the education programme ended. By contrast, participants in the video group learned about proper use of body mechanics from the "Body Mechanics Educational Video for LDH Patients" presented on a laptop, after which we also answered any questions that participants asked. Video-based education took nearly 15 min, and we provided CD-ROM with the video to the participants. Unlike participants in the intervention groups, ones in the control group did not receive structured education. Clinical nurses orally informed them about points to consider while performing activities such as standing, rising from bed and lifting. Final data collection took place in the sixth postoperative week, following the statement of the American Association of Neuroscience Nurses that pain and disability begin to decrease and that quality of life begins to increase 4-6 weeks after thoracolumbar surgery (Starkweather et al., 2013). During the postoperative period, participants in all groups completed the SF-MPQ, the ODI and the Physical Functioning and Bodily Pain subscales of the SF-36. Participants in the brochure and video groups also completed the survey addressing their satisfaction with the educational materials, whereas ones in the control group completed the survey addressing their satisfaction with the clinical education that they received. We collected data face-to-face with participants, which took approximately 20 min. Participants who lived outside Ankara completed the respective survey via telephone interviews, which took approximately 30 min.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised in preparation to receive LDH surgery and who volunteered to participate
* Older than 18 years
* Could read and write in Turkish
* Scored between 1 and 3 in the classification systems of the American Society of Anesthesiologists were preparing for their first LDH surgical operation
* Could use CD-based educational materials

Exclusion Criteria:

* Patients hospitalised in preparation to receive LDH surgery and who unvolunteered to participate
* All potential participants who had previously undergone LDH surgery
* Could not use CD-based educational materials or had mental disorders liable to prevent communication

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Subscales of the Medical Outcomes Study Short-Form 36-Item Health Survey (SF-36) | Change from quality of life at 6 weeks
  Of the instrument's eight subscales and 36 items, we used the Physical Functioning (i.e. 10 items) and Bodily Pain (i.e. 2 items) subscales. Final scores for each subscale are calculated by dividing the score obtained by the number of items on the subscale. Final scores on the subscales range from 0 to 100; higher scores indicate higher quality of life
Oswestry Disability Index (ODI) | Change from disability at 6 weeks
  The ODI has 10 questions addressing the intensity of pain, personal care, walking, sitting, standing and lifting behaviours, sex life, social life, sleep routines and travelling tendencies. Patients respond to each question on a 6-point Likert scale; for each question, scores range from 0 (i.e. no disability) to 5 (i.e. most severe disability). By contrast, total scores range between 0 and 50 and are interpreted to indicate minimal disability (0-4 points), moderate disability (5-14 points), severe disability (15-24 points), crippled (25-34 points) or bed-bound (35-50 points)
Short-Form McGill Pain Questionnaire (SF-MPQ) | Change from pain at 6 weeks
  This questionnaire evaluated the reliability and validity of the Turkish version of the instrument. The scale evaluates acute pain and consists of sensory, affective and intensity subscales; higher scores indicate a higher intensity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Özgü Bakçek, Principal Investigator — Health Science University Gulhane Faculty of Nursing, ANKARA
Locations (1):
- Özgü Bakçek, Ankara, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the study publish, we actually shared all procedurs.
Supporting Information: Study Protocol
Time Frame: Data collection have been completed